CLINICAL TRIAL: NCT05725382
Title: Can Nociception Level-guided Remifentanil Dosing Reduce Postoperative Pain in Children During General Anesthesia: A Blinded, Randomized Controlled Trial
Brief Title: Nociception Level-guided Remifentanil Dosing in Children During General Anesthesia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Pia Jaeger, MD, PhD (Other)
Responsible Party: Sponsor-Investigator, Pia Jaeger, MD, PhD, Senior Registrar, Rigshospitalet, Denmark
Organization: Rigshospitalet, Denmark (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NOL1-2022
Record Dates: First submitted 2023-01-26; First posted 2023-02-13 (Actual); Last update posted 2023-08-24 (Actual); Status verified 2023-08

CONDITIONS: Surgical Procedure, Unspecified
Keywords: Pediatric; Pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Intervention Model Description: Blinded, randomized, controlled multicenter trial with two parallel groups and a superiority design.
Who Masked: Participant, Outcomes Assessor
Masking Description: The patients and their relatives, outcome assessors, data analysts and PACU nurses will be blinded. However, the anesthesiologists and anesthesia nurses anesthetizing the child according to the NOL monitor/standard care cannot be blinded. The anesthesiologist and anesthesia nurses anesthetizing the child will not be involved in patient care after the patient leaves the theatre, nor in any clinical assessments, data collection or interpretation of adverse events.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NOL-guided remifentanil dosing (Experimental): Remifentanil dosing will preferentially be guided by the NOL index, but blood pressure and heart rate will be monitored and considered concurrently.
  * If the NOL index is > 25, remifentanil infusion will be increased.
  * If the NOL index is < 10 the remifentanil infusion rate will be reduced
  Interventions: Device: The NOL monitor (Pain Monitoring Device monitor-PMD200™)
- Standard care remifentanil dosing (No Intervention): Remifentanil dosing will be administered according to standard care per institutional practice.

INTERVENTIONS:
Device: The NOL monitor (Pain Monitoring Device monitor-PMD200™) — NOL-guided perioperative remifentanil administration
  Other Names: NOL-guided remifentanil dosing
  Arms: NOL-guided remifentanil dosing

SUMMARY:
The investigators aim to investigate whether administration of a short-acting opioid (remifentanil) guided by a pain monitor (nociceptive level monitor) during anesthesia, can reduce pain in children after surgery.

The investigators hypothesize that pain monitor-guided administration of remifentanil can reduce pain postoperatively compared with standard care.

DETAILED DESCRIPTION:
NOL-guided analgesia has not previously been assessed in children, and it is unknown whether this additional monitoring has any clinical benefits in a pediatric population.

In the present study the investigators aim to investigate whether administration of perioperative remifentanil guided by the CE-certified Pain Monitoring Device monitor-PMD200™, also called NOL-monitor, can reduce pain (primary endpoint), opioid consumption and agitation in children aged 3-16 years undergoing surgery with intravenous anesthesia.

The investigators hypothesize that NOL-guided perioperative remifentanil administration can reduce postoperative pain compared with standard clinical care (remifentanil dosing based on hemodynamic variables).

All patients will receive standard analgesia and antiemetic administered perioperatively:

* IV paracetamol 15 mg/kg
* IV Ibuprofen 10 mg/kg, unless contraindicated
* IV Morphine 25-100 μg/kg according to the extent of surgery and the departments' standard, administered 30 minutes before end of surgery (will not be included in the total perioperative or postoperative opioid consumption)
* In case of minor surgery, 1-2 μg/kg fentanyl, according to the department's standard, may be administered instead of morphine at the discretion of the anesthetist (will not be included in the total perioperative or postoperative opioid consumption)
* Regional anesthesia may be provided at the discretion of the anesthetist
* IV ondansetron 100 μg/kg

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiology (ASA) class of 1-3
* Scheduled surgery requiring intraoperative opioid administration
* Planned maintenance anesthesia with propofol and remifentanil
* The trial subject's custody holders' must be able to understand the trial protocol, risks, and benefits, and provide signed informed consent

Exclusion Criteria:

* Inability of the trial subject's custody holder to read or write Danish
* Children who cannot cooperate to the study assessments based on the investigators' evaluation. This may be children with mental disorders, visual disturbances, hearing or speech impairment etc. interfering with assessments.
* Arrythmias, either known arrythmias preoperatively or arrythmias detected within the first minutes perioperatively (in which case the patient will be excluded post- randomization).
* Allergy to the medicines used in the study
* Daily intake of opioids (morphine, oxycodone, ketobemidone, methadone, fentanyl) during the last 4 weeks
* Weight < 10 kg

Ages: 3 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 264 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2025-10-30 (Estimated); Study Completion 2025-11-01 (Estimated)

PRIMARY OUTCOMES:
First pain score assessed at the PACU | Assessed at the first time the child is awake at the PACU
  Pain at rest assessed using the Faces Pain Scale - Revised (0-100 mm).

SECONDARY OUTCOMES:
Opioid consumption at the PACU | From extubation until discharge from PACU
  Total, cumulative, opioid consumption, calculated as IV fentanyl equivalents
Perioperative opioid consumption | From induction until extubation
  Total, cumulative, perioperative opioid consumption, calculated as IV remifentanil equivalents. The planned administration of morphine/fentanyl at the end of surgery will NOT be included.
Opioid consumption after discharge from PACU and until the 48-h anesthesia followup | From PACU discharge and until the 48-hours anesthesia followup
  Total, cumulative, opioid consumption, calculated as IV morphine equivalents
Faces Pain Scale - Revised scores at rest during the PACU stay | Assessed at 15, 30, 45 and 60 minutes after arrival at the PACU, and thereafter every 30 minutes until discharge.
  Pain at rest, assessed using the Faces Pain Scale - Revised (Revised (0-100 mm), calculated as the area under the curve. If the child is sleeping, a pain score of 0 will be assigned.
FLACC pain scores at rest during the PACU stay | Assessed at 15, 30, 45 and 60 minutes after arrival at the PACU, and thereafter every 30 minutes until discharge.
  Pain at rest assessed using the Face Legs, Activity, Cry and Consolability scale (FLACC, 0-10 points), calculated as area under the curve.
Postoperative agitation | Assessed at 15, 30, 45 and 60 minutes after arrival at the PACU, and thereafter every 30 minutes until discharge.
  Postoperative agitation assessed using the WATCHA scale (0-4). The highest score at any time point will be used for the comparison between groups.

OTHER OUTCOMES:
PACU length of stay. | Assessed as time from extubation (in case there is a wait for a PACU bay) and until PACU discharge readiness, defined as the time the participant fulfils local discharge criteria
  PACU length of stay.
Postoperative nausea or vomiting | Will be assessed twice; 1) at the PACU and 2) from PACU discharge and until the 48-hour follow up.
  Assessed as a dichotomous endpoint, as either presence or absence of nausea or vomiting at any time point, during the period.
Number of events of hemodynamic instability | Perioperatively
  Number of events of hemodynamic instability requiring drug or fluid administration perioperatively.
Time to extubation | From anesthesia maintenance is stopped until the patient is extubated/LMA is removed
  The time from anesthesia maintenance is stopped until the patient is extubated/LMA is removed
Parental satisfaction. | Assessed at 48 hours postoperatively, for the entire period 0-48 hours postoperatively
  Parental satisfaction with anesthesia assessed on a numeric rating scale from 0 to 10.
Time where the NOL index value is > 25 | From the start of induction and until the time of extubation
  Time (minutes) where the NOL index value is > 25
Maximum NOL index | From the start of induction and until the time of extubation
  The highest NOL index during a 5-minute period at any time perioperatively
Mean NOL index | From the start of induction and until the time of extubation
  The mean NOL index during surgery

CONTACTS AND LOCATIONS:
Overall Officials: Pia Jæger, MD, PhD, Study Chair — Department of Anaesthesia, The Juliane Marie Center, Rigshospitalet
Locations (4):
- Denmark (4):
  - Department of Anaesthesia, The Center of Head and Orthopaedics, Rigshospitalet, Copenhagen
  - Department of Anaesthesia, The Juliane Marie Center, Copenhagen University Hospital, Rigshospitalet, Copenhagen
  - Department of Anaesthesia, Sjællands Universitetshospital, Køge, Køge
  - Department of Anaesthesia, Vejle Sygehus, Vejle